CLINICAL TRIAL: NCT00299208
Title: Phase II, Open Label, Randomized Study of Azithromycin Combination Therapy for the Treatment of Acute, Uncomplicated Falciparum Malaria
Brief Title: Azithromycin Combination Therapy for Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-149; A0661129
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-03

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Artesunate; Azithromycin; Quinine

INTERVENTIONS:
Drug: Artesunate
Drug: Azithromycin
Drug: Quinine

SUMMARY:
The goal of this study is to develop a safe, well tolerated, and highly efficacious azithromycin combination treatment for uncomplicated falciparum malaria. Azithromycin is a drug that has shown potential for malaria treatment. It will be combined with other malaria drugs currently approved for treatment in Thailand. About 120 people, ages 20-65, will be enrolled in Thailand. Participants will have severe cases of malaria and they will be hospitalized 28 days for treatment.

DETAILED DESCRIPTION:
The study is aimed at identifying a well tolerated, practical and highly efficacious treatment regimen of azithromycin in combination with artesunate or quinine for uncomplicated falciparum malaria for future studies, to monitor for the tolerability and safety of these combination regimens and to compare tolerability, safety and efficacy of azithromycin when given in combination with artesunate as compared to quinine. This study is also aimed at comparing tolerability, safety and efficacy of the combination of artesunate and azithromycin when given as a single daily dose (200mg As+1000mg Az) for 3 days as compared to 2 doses of 100mg As+750mg Az per day for 3 days and to compare the tolerability, safety and efficacy of the combination of quinine and azithromycin when given as 3 daily doses of quinine (10mg/kg) + Az 500mg vs. 2 daily doses of quinine (10mg/kg) + Az 750mg when given for 3 days.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic falciparum malaria infection as determined by malaria smear with a parasite density of 100 to 100,000 asexual parasites/µL with fever, defined as >37.5ºC, during the current illness, or history (within the last 48 hours) of fever.
2. Age: 20-65 years old
3. Male or female. All females are required to have a negative human chorionic gonadotropic (hCG) pregnancy test (urine). All females of childbearing potential (not surgically sterile, or less than two years post menopausal) are required to use an acceptable method of contraception, such as implant, injectable, oral contraceptive(s) with additional barrier contraception, intrauterine device, sexual abstinence, or vasectomized partner, throughout the study.
4. Written informed consent obtained.
5. Willing to stay hospitalized for 28 days for treatment and observations.
6. Otherwise healthy outpatients (with no other clinically-significant illnesses as described in Exclusion Criteria, #6).

Exclusion Criteria:

1. Pregnant women, nursing mothers, or women of childbearing potential who do not use an acceptable method of contraception (as described in Inclusion Criteria, #3).
2. Mixed malaria infection on admission by malaria smear.
3. A previous state of intolerance or hypersensitivity to the study drugs quinine, artesunate, or azithromycin or to drugs with similar chemical structures (quinidine, any artemisinin derivative, and macrolides such as erythromycin).
4. Malaria drug therapy administered in the past 30 days by history (quinine, chloroquine, mefloquine, artemisinin derivatives, sulfadoxine/pyrimethamine, lumefantrine).
5. Previous participation in this trial, or participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study.
6. Clinically significant illness (intercurrent illness e.g. pneumonia, pre-existing condition e..g. malignancy or conditions that may effect absorption of study medication e.g. severe diarrhea or any signs of malnutrition as defined clinically).
7. Laboratory evidence or history of significant cardiovascular, liver or renal functional abnormality, which in the opinion of the investigator would place them at increased risk. Specifically, the following will serve as exclusionary laboratory values:

   1. Creatinine > 1.4 X ULN (>2.0 mg/dl),
   2. Glucose < LLN (75 mg/dl),
   3. AST, ALT > 3x ULN (120 U/L), or
   4. Prolonged QT wave on baseline electrocardiogram (QT >0.45s)
8. Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
9. Signs or symptoms of severe malaria.
10. Anyone who received a transfusion of red blood cells within the prior 30 days.
11. Unable and/or unlikely to comprehend and/or follow the protocol.
12. Self-reported alcohol and/or any other drug abuse.
13. Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University Hospital for Tropical Diseases, Bangkok, Thailand